CLINICAL TRIAL: NCT03256851
Title: Telephone-Delivered Interventions to Target Multiple Sclerosis Fatigue
Brief Title: Telephone-Delivered Exercise for Multiple Sclerosis Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Multiple Sclerosis Society (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Nora Fritz, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1612000180
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis; Fatigue; Physical Activity
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Delivered Exercise (Active Comparator): Participants in the in-person training group will:
  1. participate in a home exercise program including aerobic training 2x/week and strength training 3x/week.
  2. complete one of their prescribed training sessions (lasting 1 hour total) each week with a physical therapist or trained member of the research team. Training sessions will focus on progression of aerobic and strength training exercises.
  Interventions: Behavioral: In-Person Delivered Exercise Therapy
- Telephone-Delivered Exercise (Experimental): Participants in the telephone-delivered training group will:
  1. participate in a home exercise program including aerobic training 2x/week and strength training 3x/week.
  2. receive a 60-minute, 1x/week telephone call from a trained research team member. Participants will report their progress from the prior week, discuss/troubleshoot any issues or problems, and receive progressions of both aerobic and strength training exercises for the upcoming week.
  Interventions: Behavioral: Telephone-Delivered Exercise Therapy

INTERVENTIONS:
Behavioral: Telephone-Delivered Exercise Therapy — A combination of aerobic and resistance training has been shown to be most effective for reducing fatigue in persons with MS.
  Aerobic training will consist of: 30 minutes of either cycling, treadmill walking or overground walking, 2x/week. Participants will be given a wrist-worn pedometer with heart-rate monitor to track their heart rate during training. Participants will be progressed to reach 60-70% of their maximal heart rate during aerobic training over the course of the study.
  Strength training will consist of hip extension, hip flexion, hip abduction, knee extension and knee flexion movements with resistance bands performed 3x/week.
  This home exercise program will be paired with a 1x/week telephone call with an investigator.
  Arms: Telephone-Delivered Exercise
Behavioral: In-Person Delivered Exercise Therapy — A combination of aerobic and resistance training has been shown to be most effective for reducing fatigue in persons with MS.
  Aerobic training will consist of: 30 minutes of either cycling, treadmill walking or overground walking, 2x/week. Participants will be given a wrist-worn pedometer with heart-rate monitor to track their heart rate during training. Participants will be progressed to reach 60-70% of their maximal heart rate during aerobic training over the course of the study.
  Strength training will consist of hip extension, hip flexion, hip abduction, knee extension and knee flexion movements with resistance bands performed 3x/week.
  This home exercise program will be paired with a 1x/week visit to the laboratory to work with a physical therapist or trained team member.
  Arms: In-Person Delivered Exercise

SUMMARY:
Multiple sclerosis (MS) is a progressive demyelinating disorder that damages white matter in the central nervous system. Although individuals experience mobility (e.g., walking, balance) impairments that lower quality of life and limit participation in daily activities, one of the most prominent symptoms is fatigue. Up to 92% of individuals report fatigue that manifests as lack of energy, exhaustion or worsening of MS symptoms and ultimately contributes to increasing disability. The currently available pharmaceutical treatments fail to fully control fatigue in the majority of individuals with MS; non-pharmacologic therapies such as exercise and behavioral therapies offer the best hope for combating MS fatigue in the majority of individuals.

Exercise therapy is effective in reducing MS fatigue. However, access to exercise therapy is seriously limited for many individuals with MS due to geographical location, limited resources (e.g., financial, transportation), and/or disability. Thus, the development and evaluation of an alternative delivery method for exercise therapy to target MS-related fatigue that increases participation and reduces barriers is critical.

In this study, the investigators will compare traditional in-person delivered exercise therapy to telephone-delivered exercise therapy to target fatigue in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS, SPMS, or PPMS
* Ambulatory for at least 5 minutes at a time
* Self-reported fatigue on Fatigue Severity Scale
* Able to follow study-related commands
* Able to attend study appointments

Exclusion Criteria:

* MS exacerbation within the past 30 days
* Evidence of another neurological disorder or orthopedic disorder that would interfere with exercise participation
* Acute illness or injury that prevents participation in the intervention
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kratz AL, Atalla M, Whibley D, Myles A, Thurston T, Fritz NE. Calling Out MS Fatigue: Feasibility and Preliminary Effects of a Pilot Randomized Telephone-Delivered Exercise Intervention for Multiple Sclerosis Fatigue. J Neurol Phys Ther. 2020 Jan;44(1):23-31. doi: 10.1097/NPT.0000000000000296. PMID 31738192

RESULTS

PARTICIPANT FLOW:
Groups:
- In-Person Delivered Exercise: Participants in the in-person training group will:
  1. participate in a home exercise program including aerobic training 2x/week and strength training 3x/week.
  2. complete one of their prescribed training sessions (lasting 1 hour total) each week with a physical therapist or trained member of the research team. Training sessions will focus on progression of aerobic and strength training exercises.
  In-Person Delivered Exercise Therapy: A combination of aerobic and resistance training has been shown to be most effective for reducing fatigue in persons with MS.
  Aerobic training will consist of: 30 minutes of either cycling, treadmill walking or overground walking, 2x/week. Participants will be progressed to reach 60-70% of their maximal heart rate during aerobic training over the course of the study.
  Strength training will consist of hip extension, hip flexion, hip abduction, knee extension and knee flexion movements with resistance bands performed 3x/week.
- Telephone-Delivered Exercise: Participants in the telephone-delivered training group will:
  1. participate in a home exercise program including aerobic training 2x/week and strength training 3x/week.
  2. receive a 60-minute, 1x/week telephone call from a trained research team member. Participants will report progress from the prior week, troubleshoot any issues, and receive progressions of both aerobic and strength exercises for the upcoming week.
  Telephone-Delivered Exercise Therapy: A combination of aerobic and resistance training has been shown to be most effective for reducing fatigue in persons with MS.
  Aerobic training will consist of: 30 minutes of either cycling, treadmill walking or overground walking, 2x/week. Participants will be progressed to reach 60-70% of their maximal heart rate during aerobic training over the course of the study.
  Strength training will consist of hip extension, hip flexion, hip abduction, knee extension and knee flexion movements with resistance bands performed 3x/week.
Period: Overall Study
Arm/Group | In-Person Delivered Exercise | Telephone-Delivered Exercise
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Person Delivered Exercise | Telephone-Delivered Exercise | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (7.4) | 45.9 (8.0) | 48.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
Fatigue Severity Scale [Mean (Standard Deviation); unit: units on a scale] — The Fatigue Severity Scale is a 9-item questionnaire in which participants rate their fatigue from 1-7 for each question. A higher score (max total = 63) indicates worse fatigue.
  The total score is reported. The range of possible scores is 9-63.
  units on a scale | 51.1 (4.1) | 47.8 (9.5) | 48.5 (7.3)
Patient Determined Disease Steps (PDDS) [Mean (Inter-Quartile Range); unit: units on a scale] — The PDDS requires a single response on a 0-8 scale that indicates the person's perceived level of disability from 0 (normal - I have some mild symptoms, mostly sensory due to MS but they do not limit my activity) to 8 (bedridden- unable to sit in a wheelchair for more than one hour).
  The total score is reported, with higher numbers indicating worse disability.
  units on a scale | 3.5 [3 to 5] | 2 [1 to 3] | 3 [1 to 4]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.1 [27.1 to 34.7] | 33.8 [30.8 to 38.7] | 32.9 [27.8 to 36.4]
Years Since Diagnosis [Median (Inter-Quartile Range); unit: years] | 4.5 [4 to 9] | 13.5 [5 to 16] | 8 [4 to 13.5]

OUTCOME MEASURES:

1. Primary Outcome: Daily Average Fatigue Intensity Score
Description: Rated on a 0-10 numerical rating scale, entered directly on the PRO-Diary (CamNTech, Cambridge, UK), which provides a more reliable and sensitive assay of symptoms compared to traditional recall measures.
  A score of 0 indicates no fatigue and a score of 10 indicates extremely severe fatigue.
Time Frame: Baseline (pre) and 8 weeks (post)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Person Delivered Exercise | Telephone-Delivered Exercise
Number analyzed (Participants) | 9 | 10
units on a scale
  Pre | 3.9 (1.9) | 4.4 (1.1)
  Post | 3.2 (1.9) | 2.3 (1.5)

2. Primary Outcome: Daily Average Fatigue Interference Score
Description: Rated on a 0-10 numerical rating scale, entered directly on the PRO-Diary (CamNTech, Cambridge, UK), which provides a more reliable and sensitive assay of symptoms compared to traditional recall measures.' A score of 0 indicates no interference while a score of 10 indicates complete interference (i.e., worse).
Time Frame: Baseline (pre) and 8 weeks (post)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Person Delivered Exercise | Telephone-Delivered Exercise
Number analyzed (Participants) | 9 | 10
units on a scale
  Pre | 3.1 (1.9) | 3.0 (1.3)
  Post | 2.7 (1.8) | 1.5 (1.7)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | In-Person Delivered Exercise | Telephone-Delivered Exercise
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03256851/Prot_SAP_000.pdf